CLINICAL TRIAL: NCT01358188
Title: Prospective Study of Macrophage Activation and Cross Talk Between Immune System Elements in Subjects With Gaucher Disease
Brief Title: Exploration of Immunity in Gaucher Disease
Status: Completed | Type: Observational
Sponsor: O & O Alpan LLC (Other)
Responsible Party: Principal Investigator, Ozlem Goker-Alpan, MD, Chief Medical Officer, O & O Alpan LLC
Other Study IDs: 10-CFCT-01
Record Dates: First submitted 2011-05-06; First posted 2011-05-23 (Estimated); Last update posted 2017-04-04 (Actual); Status verified 2017-04

CONDITIONS: Gaucher Disease
Keywords: Gaucher disease; immunity; inflammation; macrophage activation
MeSH Terms: conditions — Gaucher Disease; Inflammation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Gaucher disease group: Subjects will include individuals with GD
- Control group: Controls will include healthy individuals and individuals with primary immune dysfunction

SUMMARY:
Gaucher disease (GD), the inherited deficiency of the lysosomal enzyme glucocerebrosidase is characterized with accumulation of abnormal lipid in cells of the immune system, called macrophages. Lipid engorged macrophages, then become activated, and are also called "Gaucher cells". The mechanisms leading to macrophage activation is not fully known, however several findings in individuals with GD, such as non-specific inflammation,clinically resembling a rheumatic disease with an increased sedimentation rate, joint pain, and extreme fatigue, in addition poor wound healing, and a predisposition to diabetes may suggest an inappropriately functioning immune system in GD. The pathways leading to macrophage activation could be related to the accumulation of lipid metabolites or through the effects of other immune cells. In this study, immunologic profiling and functional assays will be performed in peripheral blood samples from patients with GD. The identification of the immunologic basis of GD will lead to the the development of new disease markers and different treatment options.

DETAILED DESCRIPTION:
Activated lipid engorged macrophages are the hallmark for Gaucher disease (GD). The evidence for this activation comes from the clinical finding of 1000-fold increase of serum chitotriosidase, a chitinase specifically secreted from activated macrophages. While these markers decrease with the initiation of therapy, they are not specific for organ involvement. The mechanisms of this macrophage activation is unclear, however, the presence of a non-specific inflammatory response (e.g. high sedimentation rate), poor wound healing and insulin resistance in Gaucher patients point to its clinical relevance. The finding of T, B and NK cell abnormalities in Gaucher patients also suggest either direct effects of GD lipid metabolites or indirect mechanisms via macrophages. Therefore, understanding the mechanisms of macrophage activation and the crosstalk with other immune cell types could provide mechanistic insights for pathogenesis of GD.

The investigators hypothesize that in GD the mechanisms leading macrophage activation could be related either directly to the accumulation of the lipid metabolites or through the effects of other cells of the immune system. To determine the pathways leading to macrophage dysregulation in GD, the investigators will evaluate the functional response of monocytes isolated from GD patients and profile of T cell and NK cell subsets in peripheral blood of these patients. The investigators will then assess whether macrophage dysfunction in GD is caused by an primary alteration immune response (NK and T cells response) or secondary due to the direct effects of substrate accumulation performing immunological profiling of GD patient blood samples, and through functional assays. Identification of the immunological basis of GD pathogenesis could lead to the development of both biomarkers and novel approaches for therapeutic interventions to alleviate disease symptoms. In addition, our studies will reveal novel effects of the accumulation of the lipid substrate in GD in modulating macrophage and lymphocyte subsets.

ELIGIBILITY:
Inclusion Criteria:

* History of Gaucher disease
* Nonspecific inflammatory response evidenced by an increased ESR or positive CRP
* Positive markers for autoimmune disorders such as ANA, RF
* Chronic inflammatory disorders such as inflammatory bowel disease
* NIDDM
* Otherwise would qualify for an immunological work-up such as opportunistic or unusual infections such as atypical mycobacterial infections, unexplained lymphadenopathy.

Exclusion Criteria:

* Severe cognitive deficits impairing decision making
* Pregnant or nursing, as these conditions may alter immunologic profile
* History of Hepatitis B, C or HIV infections

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study population will include individuals with Gaucher disease, healthy controls and individuals with primary immune dysfunction
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2011-04; Primary Completion 2016-05-02 (Actual); Study Completion 2016-05-02 (Actual)

PRIMARY OUTCOMES:
Macrophages from patients with GD and primary immune hypo/dysfunction will show higher level of activation markers. | 2 years
  The effect of macrophage activation on inflammation and immune response in subjects GD:
  As measured by 1) The secretion of proinflammatory cytokines/chemokines ( IL-1b, TNF, IL-6 and Mip1a ) 2) The ability of macrophages to shape the differentiation profile of naïve and memory T cells.

CONTACTS AND LOCATIONS:
Overall Officials: Ozlem Goker-Alpan, M.D., Principal Investigator — Center for Clinical Trials, O&O Alpan
Locations (1):
- Lysosomal Diseases Research and Treatment Center, CFCT, Fairfax, Virginia, United States

REFERENCES:
- [Background] Goker-Alpan O. Optimal therapy in Gaucher disease. Ther Clin Risk Manag. 2010 Jul 21;6:315-23. doi: 10.2147/tcrm.s6955. PMID 20668714